CLINICAL TRIAL: NCT00963300
Title: Hypoxia Assessment in Localized Prostate Cancer: A Companion Protocol to a Phase II Study of Stereotactic Body Radiation Therapy (SBRT) for Low and Intermediate Risk Prostate Cancer
Brief Title: MRI in Assessing Hypoxia in Patients With Localized Prostate Cancer Undergoing Stereotactic Body Radiation Therapy
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Project Never Initiated - no human subjects were enrolled and no data regarding humans was collected or studied
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SCCC-062009-014; CDR0000652306 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2009-08-20; First posted 2009-08-21 (Estimated); Last update posted 2018-11-26 (Actual); Status verified 2018-11

CONDITIONS: Prostate Cancer
Keywords: adenocarcinoma of the prostate; stage I prostate cancer; stage IIB prostate cancer; stage IIA prostate cancer; stage III prostate cancer; stage IV prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Magnetic Resonance Spectroscopy

INTERVENTIONS:
Procedure: blood-oxygen-level-dependent functional magnetic resonance imaging
Procedure: dynamic contrast-enhanced magnetic resonance imaging
Procedure: magnetic resonance spectroscopic imaging
Procedure: tissue-oxygen-level-dependent functional magnetic resonance imaging

SUMMARY:
RATIONALE: Diagnostic procedures, such as MRI, may help measure oxygen levels in tumor cells. It may also help doctors predict a patient's response to treatment and help plan the best treatment.

PURPOSE: This clinical trial is studying how well MRI works in assessing hypoxia in patients with localized prostate cancer undergoing stereotactic body radiation therapy.

DETAILED DESCRIPTION:
OBJECTIVES:

* To characterize the status of global hypoxia within the prostate before stereotactic body radiotherapy (SBRT) as assessed by blood-oxygen-level-dependent and tissue-oxygen-level-dependent MRI.
* To characterize tumor vasculature and metabolism within the prostate before SBRT as assessed by dynamic contrast-enhanced MRI and magnetic resonance spectroscopic imaging, respectively.
* Correlate prostate and normal tissue hypoxia before SBRT with clinical outcomes (toxicity and biochemical [PSA] control) after SBRT.

OUTLINE: Within 1-3 weeks before beginning stereotactic body radiotherapy, patients undergo T2-weighted anatomic MRI, magnetic resonance spectroscopic imaging, blood-oxygen-level-dependent and tissue-oxygen-level-dependent MRI, and dynamic contrast-enhanced MRI.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Biopsy proven adenocarcinoma of the prostate

  * Localized disease
* Scheduled to undergo treatment with stereotactic body radiotherapy (SBRT) on a phase II clinical trial

  * Has not yet started SBRT

PATIENT CHARACTERISTICS:

* Serum creatinine ≤ 1.2 mg/dL
* No claustrophobia
* No other contraindication to MRI (e.g., implanted pacemaker device)
* No known allergy to MRI contrast

PRIOR CONCURRENT THERAPY:

* No prior treatment for prostate cancer (e.g., hormonal therapy or chemotherapy)

Ages: 18 Years to 120 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-09 (Estimated); Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Status of global hypoxia within the prostate as assessed by blood-oxygen-level-dependent and tissue-oxygen-level-dependent MRI
Tumor vasculature and metabolism within the prostate as assessed by dynamic contrast-enhanced MRI and magnetic resonance spectroscopic imaging
Correlation of prostate and normal tissue hypoxia before treatment with clinical outcomes after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Robert D. Timmerman, MD, Principal Investigator — Simmons Cancer Center